CLINICAL TRIAL: NCT06454539
Title: The Effect of Functional Inspiratory Muscle Training Versus Inspiratory Muscle Training on Trunk Control and Respiratory Functions in Patients With Chronic Stroke
Brief Title: The Effect of Functional Inspiratory Muscle Training Versus Inspiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2024-06-02; First posted 2024-06-12 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Muscles; Stroke
Keywords: Inspiratory Muscles Training; Exercise; Chronic Stroke; Neurodevelopmental Treatment
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-IMT Group (Experimental): Participants in this group will apply functional IMT as a supervised program 3 days a week, and IMT as a home program on 2 different days. In functional IMT, participants will perform breathing exercises with the device while simultaneously performing exercises based on the neurodevelopmental treatment approach given below.
  Interventions: Other: Functional Inspiratory Muscle Training
- IMT Group (Active Comparator): Participants in this group will perform supervised neurodevelopmental treatment approach-based exercises and IMT 3 days a week, and IMT as a home program on 2 different days.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training — Functional IMT is an inspiratory muscle training that ensures core stabilization and maintains postural control. Rhythmic co-contractions of the core muscle areas (diaphragm, transversus abdominis, multifidus, pelvic floor) ensure the stability of the trunk and provide it with the feature of being the support point of movement. In the first stage, the person is given core stabilization training. Secondly, core stabilization is maintained and continued with strong trunk activation exercises. Postural exercises reinforce the other function of the breathing muscles, which is actually 'core' stabilization.
  Arms: F-IMT Group
Other: Inspiratory Muscle Training — Inspiratory muscle training (IMT) is one of the methods used to increase respiratory muscle strength. Different tools and methods (threshold resistive loading, normocapnic hyperpnea, and threshold pressure loading) have been developed for IMI. The most used method in the literature is the threshold pressure loading method. This method requires subjects to generate a negative pressure sufficient to overcome the load of the device and thus initiate inspiration. ICE is most commonly performed in a sitting position, with upper extremities supported and upper chest/shoulders relaxed. By placing the person in this position, the aim is for the respiratory muscles to focus only on the work of breathing.
  Arms: IMT Group

SUMMARY:
This study aims to compare the effectiveness of functional inspiratory muscle training (IMT) versus inspiratory muscle training on trunk control, respiratory parameters, activity, and participation in chronic stroke patients. The study is a prospective, randomized, and parallel study. Forty-four stroke patients who meet the inclusion and exclusion criteria will be included in the study. The patients to be included in the study will be divided into equal numbers into two groups, F-IMT Group, and IMT Group, by block randomization method. Participants' trunk control will be measured with the Trunk Disability Scale and Trunk Control Test, respiratory parameters will be measured with respiratory muscle strength measurement test and respiratory function test, balance and gait will be measured with the Berg Balance Scale, and core muscle will be measured with pressurized biofeedback unit, exercise capacity will be measured by 6 minutes of walking. In the test, the level of independence in daily living activities will be evaluated with the Barthel Activities of Daily Living Index and treatment satisfaction with the Global Change Scale. Participants in the Functional IMT Group will perform supervised functional IMT 3 days a week, and IMT as a home program on 2 different days. In functional IMT, participants will perform breathing exercises with the device while simultaneously performing exercises based on the neurodevelopmental treatment approach given below. Exercises will be applied progressively, taking into account the functional status of stroke patients. Participants in the IMT Group will perform supervised exercises and IMT based on a neurodevelopmental treatment approach 3 days a week, and IMT as a home program on 2 different days.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of functional inspiratory muscle training (IMT) versus inspiratory muscle training on trunk control, respiratory parameters, activity, and participation in chronic stroke patients.

For this purpose, our hypotheses were determined as follows:

H0: There is no difference between the effects of inspiratory muscle training and functional inspiratory muscle training applied in addition to the neurodevelopmental treatment approach in chronic stroke patients on trunk control, respiratory muscle strength, respiratory parameters, walking, balance, core muscles, functional capacity, daily living activities, and exercise adaptation.

H1: There is a difference between the effects of inspiratory muscle training and functional inspiratory muscle training applied in addition to the neurodevelopmental treatment approach in chronic stroke patients on trunk control, respiratory muscle strength, respiratory parameters, walking, balance, core muscles, functional capacity, daily living activities and exercise adaptation. has.

The study is a prospective, randomized, and parallel study. Forty-four stroke patients who meet the inclusion and exclusion criteria will be included in the study. The patients to be included in the study will be divided into equal numbers into two groups, F-IMT Group, and IMT Group, by block randomization method. Participants' trunk control will be measured with the Trunk Disability Scale and Trunk Control Test, respiratory parameters will be measured with respiratory muscle strength measurement test and respiratory function test, balance and gait will be measured with the Berg Balance Scale, and core muscle will be measured with pressurized biofeedback unit, exercise capacity will be measured by 6 minutes of walking. In the test, the level of independence in daily living activities will be evaluated with the Barthel Activities of Daily Living Index and treatment satisfaction with the Global Change Scale. Participants in the Functional IMT Group will perform supervised functional IMT 3 days a week, and IMT as a home program on 2 different days. In functional IMT, participants will perform breathing exercises with the device while simultaneously performing exercises based on the neurodevelopmental treatment approach given below. Exercises will be applied progressively, taking into account the functional status of stroke patients. Participants in the IMT Group will perform supervised exercises and IMT based on neurodevelopmental treatment approach 3 days a week, and IMT as a home program on 2 different days. Rehabilitation programs for stroke patients focus more on physical recovery and training on respiratory functions is kept in the background. It is expected that the inclusion of Functional IMT, an integrated exercise program that includes inspiratory muscle functions, in the rehabilitation programs of stroke patients will contribute to closing this gap. The unique value of our study is that it is conducted in stroke patients and compares the effects of Functional IMT and IMT.

In light of the data obtained from the study, it is expected that Functional IMT can be used by physiotherapists in the clinic and will contribute to other possible research.

ELIGIBILITY:
Inclusion Criteria:

Must have been diagnosed with unilateral cerebral lesions Must be able to have been diagnosed with a stroke at least 6 months ago Must be able to the mini-mental test result is more than 24 points Having a score of 3 or above on the functional ambulation scale Must be able to follow instructions and participate in work procedures Must be able to give informed consent and volunteering

Exclusion Criteria:

Neurological disease and transient ischemic attack Multiple strokes Signs of increased intracranial pressure Uncontrolled hypertension (blood pressure higher than 150/90 on three or more occasions in the last 24 hours) Gastrocnemius muscle severely spasticity Myocardial infarction, angina, or acute heart failure in the last 3 months Uncontrollable chronic disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Measurement of respiratory muscle strength | Ten week
  In the evaluation of respiratory muscle strength, maximum inspiratory intraoral pressure (MIP) and maximum expiratory intraoral pressure (MEP) will be measured using a portable, electronic oral pressure measuring device, and their values will be recorded in cmH2O. Assessment of respiratory muscle strength will be measured with a portable, electronic oral pressure measurement device (Micro Medical Micro RPM, Rochester, England).
Trunk Impairment Scale | Ten week
  It is a test developed to evaluate the trunk control of stroke patients. It includes 3 subheadings that evaluate static sitting balance, dynamic sitting balance, and coordination. It includes 3 questions on static sitting balance, 10 questions on dynamic sitting balance, and 4 questions on coordination. It is scored between 0 and 23. 0 is the lowest value and 23 is the highest value and indicates good trunk control.
Trunk Control Test | Ten week
  It is a scale obtained by modifying the scoring of the first special clinical scale developed to evaluate trunk control. The scale consists of four items, each of which is evaluated over three points (0-15-25), and the total score is min;0 - max:100.
Measurement of respiratory muscle endurance | Ten week
  Patients will undergo muscle endurance testing at increasing threshold load. The test will be performed twice on the same day, 15 minutes apart. Test times will be calculated and recorded in seconds. The result value will be obtained by multiplying the test time and the pressure value corresponding to the time.

SECONDARY OUTCOMES:
PRONE test | Ten week
  A stabilizer pressures biofeedback unit will be used for this test. Before the test, he or she will be taught an eye sit and how to contract his abdominal muscles while lying face down. He/she will be placed face down on a pillow connected to a long manometer. The long lower edge of the pillow will be parallel to the cristae, placed in the lower part of the abdomen, and they will be asked to lie down with their knees straight, spine straightness and equipment, and basic filling placed. After the pressure of the manometer is set to 70 mmHg, you will be asked to hold your breath and contract your abdominal muscles. Meanwhile, the pressure of the manometer is reduced. The test will be repeated when the pressure in the manometer decreases. The retention will be recorded. The performance will be done in three repetitions and will be kept separate from the three views.
Pulmonary function test | Ten week
  In the respiratory function test, the athletes' forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), the ratio of forced expiratory volume in the first second to forced vital capacity (FEV1/FVC), and peak flow rate (PEF) will be measured with a portable spirometer. A respiratory function test will be performed with a spirometer device (Cosmed Pony FX, Italy) according to ATS/ERS criteria.
Berg Balance Scale (BDS) | Ten week
  BDS is a scale that includes 14 instructions and scores between 0 and 4 are given by observing the patient's performance for each instruction. A score of 0 is given when the patient cannot do the activity at all, while a score of 4 is given when the patient completes the activity independently. The highest score is 56, 0-20 points indicate imbalance, 21-40 points indicate acceptable balance, and 41-56 points indicate good balance. It takes between 10 and 20 minutes to complete the scale.
Six Minute Walk Test (6MWT) | Ten week
  6MWT, which is highly reliable in stroke patients, is performed in a corridor that is at least 30 m long, has a flat and hard floor, and is marked every three meters. Turning zones should be determined by an object such as a colored traffic cone. The start and finish line are determined. The patient is asked to walk the longest distance he can in 6 minutes. The distance walked is measured and recorded.
Barthel Index for Activities of Daily Living (ADL) | Ten week
  ADL is a scale that evaluates all steps of daily living activities. It is used to determine the independence levels of individuals in their activities. Barthel index scores range from 0-100, 0-20 points; complete dependence, 21-61 points; advanced addiction, 62-90 points; moderate dependence, 91-99 points; mild addiction, 100 points; explains independence.
Evaluation of treatment satisfaction | One week
  The satisfaction levels of all participants in the study with the treatment they received at the end of the study will be evaluated with the "Global Rating of Change Scale (GROC). GROC is a scale on which patients determine, from their perspective, the amount of improvement or deterioration in their health status over time. There are different types of ratings in GROC. In our study, the form consisting of 7 levels in the -3 and +3 value ranges (-3: I am much worse, 0: I am the same, +3: I am completely healed) will be preferred.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunus Emre TÜTÜNEKEN, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No